CLINICAL TRIAL: NCT02130869
Title: A Pilot Study of Immunotherapy Including Haploidentical NK Cell Infusion Following CD133+ Positively-Selected Autologous Hematopoietic Stem Cells in Children With High Risk Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASCIST; NCI-2014-00275 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Neuroblastoma; Lymphoma; High-risk Tumor
Keywords: Autologous stem cell transplantation; Natural killer cells
MeSH Terms: conditions — Neuroblastoma; Lymphoma | interventions — Interleukin-2; aldesleukin; Hu14.18K322A monoclonal antibody; humanized 3F8 anti-GD2 monoclonal antibody; Busulfan; Melphalan; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Bendamustine Hydrochloride; Etoposide; Cytarabine; Carboplatin; Granulocyte Colony-Stimulating Factor; Filgrastim; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Group A: Neuroblastoma (Experimental): All participants first receive standard of care high-dose chemotherapy specific to their tumor type. Group A participants receive busulfan, melphalan, CD133+ selected autologous stem cell infusion, hu14.18K322A, IL-2, haploidentical natural killer cell infusion, G-CSF, and GM-CSF.
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Biological: CD133+ selected autologous stem cell infusion; Biological: IL-2; Biological: hu14.18K322A; Drug: Busulfan; Drug: Melphalan; Biological: GM-CSF; Device: Haploidentical natural killer cell infusion; Biological: G-CSF; Device: CliniMACS
- Group B: Lymphoma (Experimental): All participants first receive standard of care high-dose chemotherapy specific to their tumor type. Group B participants receive bendamustine, etoposide (or etoposide phosphate), cytarabine, melphalan, CD133+ selected autologous stem cell infusion, IL-2, haploidentical natural killer cell infusion, G-CSF, and GM-CSF.
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Biological: CD133+ selected autologous stem cell infusion; Biological: IL-2; Drug: Melphalan; Biological: GM-CSF; Drug: Bendamustine; Drug: Etoposide; Drug: Cytarabine; Device: Haploidentical natural killer cell infusion; Biological: G-CSF; Drug: Etoposide phosphate; Device: CliniMACS
- Group C: High-Risk Tumors (Experimental): All participants first receive standard of care high-dose chemotherapy specific to their tumor type. Group C participants receive melphalan, etoposide (or etoposide phosphate), carboplatin, CD133+ selected autologous stem cell infusion, IL-2, haploidentical natural killer cell infusion, G-CSF, and GM-CSF.
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Biological: CD133+ selected autologous stem cell infusion; Biological: IL-2; Drug: Melphalan; Biological: GM-CSF; Drug: Etoposide; Drug: Carboplatin; Device: Haploidentical natural killer cell infusion; Biological: G-CSF; Drug: Etoposide phosphate; Device: CliniMACS

INTERVENTIONS:
Biological: CD133+ selected autologous stem cell infusion — Hematopoietic stem cells will be collected from children with high-risk solid tumors. After collection, they will be immuno-magnetically selected using CD133 as a marker in efforts to reduce tumor cell contamination in the stem cell graft. After high dose chemotherapy, those selected stem cells will be infused, followed shortly thereafter by an infusion of haploidentical natural killer cells.
  Other Names: Natural killer (NK) cell infusion
Biological: IL-2 — Following infusion of haploidentical natural killer cells, interleukin-2 (IL-2) subcutaneously (SQ) will be given to support the in vivo survival of donor NK cells.
  Other Names: Interleukin-2; Aldesleukin; Proleukin(R)
Biological: hu14.18K322A — Participants with neuroblastoma (Group A) will receive hu14.18K322A intravenously (IV).
  Other Names: anti-GD2 antibody; Hu14.18K322MAB
  Arms: Group A: Neuroblastoma
Drug: Busulfan — Given IV - Group A only.
  Other Names: Busulfex(R); Myleran(R)
  Arms: Group A: Neuroblastoma
Drug: Melphalan — Given IV - All groups.
  Other Names: L-phenylalanine mustard; Phenylalanine mustard; L-PAM; L-sarcolysin
Biological: GM-CSF — Given SQ - All groups.
  Other Names: Sargramostim; Leukine(R)
Drug: Bendamustine — Given IV - Group B only.
  Other Names: Treanda®; Bendamustine hydrochloride
  Arms: Group B: Lymphoma
Drug: Etoposide — Given IV - Group B and Group C. In case of etoposide reactions, etoposide phosphate will be given.
  Other Names: VP-16; Vepesid(R)
  Arms: Group B: Lymphoma; Group C: High-Risk Tumors
Drug: Cytarabine — Given IV - Group B only.
  Other Names: ARA-C
  Arms: Group B: Lymphoma
Drug: Carboplatin — Given IV - Group C only.
  Other Names: Inorganic heavy metal coordination complex
  Arms: Group C: High-Risk Tumors
Device: Haploidentical natural killer cell infusion — NK cell product will be collected from donors using leukapheresis procedures. The autologous hematopoietic stem cell graft product will be positively selected using the investigational CliniMACS device and CD133 Microbead reagent. Following standard laboratory procedures, the NK cell product will be enumerated and assessed for viable cell content. NK cells will be infused by slow IV push over 3 to 15 minutes immediately after processing, evaluation and release testing.
  Other Names: NK cell infusion
Biological: G-CSF — Given SQ - All Groups.
  Other Names: Filgrastim; Neupogen(R)
Drug: Etoposide phosphate — In case of etoposide reactions, etoposide phosphate will be given IV. - Group B and Group C only.
  Other Names: Etopophos(R)
  Arms: Group B: Lymphoma; Group C: High-Risk Tumors
Device: CliniMACS — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest, such as CD3+ human T cells.
  Other Names: Cell Selection System

SUMMARY:
This is a pilot clinical trial investigating the addition of haploidentical natural killer cell infusion to autologous stem cell transplantation. This intervention will be evaluated in children with high-risk solid tumors for whom autologous transplantation is indicated. Natural killer cells from a haploidentical family member will be given after high dose chemotherapy and positively selected autologous stem cells. In patients with neuroblastoma, the anti-GD2 antibody hu14.18K322A will also be given. The effect on normal hematopoietic cell recovery will be evaluated and survival of children treated with this approach will be determined.

The investigators expect to enroll 36 participants. Haploidentical family members (donors) will also be recruited to provide natural killer cells.

DETAILED DESCRIPTION:
Primary Objective:

* To evaluate day +35 ANC engraftment in autologous stem cell transplantation for high risk pediatric malignancies after stem cell selection and immunotherapy.

Secondary Objectives

* To estimate incidence of relapse, disease-free survival and overall survival.
* To characterize lymphocyte and hematopoietic reconstitution in these patients.
* To describe the characteristics of the stem cell and natural killer cell grafts.
* To estimate the overall survival of patients treated without stem cell manipulation or NK cell infusion due to off therapy criteria

ELIGIBILITY:
The transplant recipient will be evaluated for eligibility at two time points during study participation. The first phase will be when the autologous stem cell product is collected. The recipient will later need to meet specific eligibility criterion at the time of the autologous stem cell infusion. The two phases and the respective criteria are described below.

Inclusion criteria for autologous stem cell collection (Phase 1 - transplant recipient):

* Less than or equal to 21 years of age.
* Malignancy at high risk of treatment failure for which autologous hematopoietic stem cell transplantation is considered within standard practice.

  * Group A: High-risk neuroblastoma
  * Group B: Recurrent or refractory Hodgkin lymphoma; recurrent or refractory non-Hodgkin lymphoma
  * Group C: High-risk, recurrent or metastatic sarcoma; recurrent or advanced stage Wilms tumor; desmoplastic small round cell tumor; metastatic or recurrent retinoblastoma, high-risk germ cell tumors, and high-risk brain tumors
* Sarcoma or Wilms tumor diagnosis (Group C) will require evaluation by physician in the St. Jude Solid Tumor Division, other than the referring physician, attesting that autologous SCT provides the prospect of direct benefit for the participant.
* Has a potentially suitable human leukocyte antigen (HLA) haploidentical donor available.
* Research participant or legal guardian/representative must be willing to give written informed consent
* Does not have any active or prior malignant or pre-malignant condition of the bone marrow, excluding metastasis of the primary malignancy.
* Has no known allergy to murine products or positive human anti-mouse antibody (HAMA).
* (Female only) Negative serum or urine pregnancy test (to be conducted within 7 days prior to enrollment).
* (Female only) Not breastfeeding.

Inclusion criteria to proceed with autologous stem cell transplantation (Phase 2 - transplant recipient):

* Has a confirmed suitable HLA haploidentical donor available.
* Previously collected autologous stem cell product met the minimum collection target and minimum infusion target as described in the protocol.
* At least two weeks since receipt of any biological therapy, chemotherapy, and/or radiation therapy.
* Has recovered from all acute NCI Common Toxicity Criteria grade II-IV non-hematologic toxicities from prior therapy per the judgment of the PI.
* Shortening fraction greater than or equal to 25%.
* Creatinine clearance or glomerular filtration rate greater than or equal to 50 mL/min/1.73 m^2.
* Pulse oximetry greater than or equal to 92% on room air.
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) less than or equal to 3 times the upper limit of the institution-established normal range.
* Direct bilirubin less than or equal to 3.0 mg/dL.
* Karnofsky or Lansky performance score of greater than or equal to 50.
* Has not received a prior hematopoietic stem cell transplant within 3 months.
* Has no known allergy to murine products or positive human anti-mouse antibody (HAMA)
* (Female only) Is not pregnant (negative serum or urine pregnancy test to be conducted within 7 days prior to admission for transplant).
* (Female only) Is not breastfeeding.
* Does not meet donation eligibility requirements as outlined by 21 CFR 1271 and agency guidance.

Inclusion criteria for haploidentical NK cell donor:

* At least 18 years of age.
* Partially HLA matched family member.
* Human immunodeficiency virus (HIV) negative.
* (Female only) Is not pregnant (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment).
* (Female only) Is not breastfeeding.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10-10 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Percent of participants with positive ANC engraftment | Day 35 post transplant
  Feasibility will be determined based on ANC engraftment defined as ANC ≥500/mm^3 for 3 consecutive tests performed on different days evaluated before day 35 post-transplant. If the study is considered feasible, the ANC engraftment rate will be 100% (95% Blyth-Still-Casella (BSC) CI: 76.45%-100%) without any failure, 92% (BSC 95% CI: 65.11%-99.57%) with 1 failure, and 83% (BSC 95% CI: 55%-96.95%) with 2 failures. In addition, if more than 2 (≥ 3) on-therapy patients die due to any protocol treatment-related causes during the first 12 months post-transplant across all groups (3 deaths among 36 participants), the study will be stopped. Deaths due to treatment not specified in this protocol will not be included in evaluation of this stopping rule.

SECONDARY OUTCOMES:
Overall survival | Up to one year after transplantation
  Overall survival is defined based on any death. The Kaplan-Meier Estimate will be provided.
Disease-free survival | Up to one year after transplantation
  Disease-free survival is defined based on any death, graft failure, or relapsed/resistant disease. The Kaplan-Meier Estimate will be provided.
Incidence of relapse | Up to one year after transplantation
  Cumulative incidence of relapse will be estimated using Kalbfleisch-Prentice method. Death is the competing risk event.
Lymphocyte and hematopoietic reconstitution | Up to one year after transplantation
  The hematopoietic cell recovery and engraftment rates will be reported with a Blyth-Still-Casella 95% confidence interval.
Characteristics of the stem cell grafts | Up to one year after transplantation
  Results will be reported and presented descriptively.
Characteristics of the natural killer cell grafts. | Up to one year after transplantation
  Results will be reported and presented descriptively.
Overall survival of patients treated without stem cell manipulation or NK cell infusion due to off therapy criteria | Up to one year after transplantation
  The Kaplan-Meier estimate will be provided for overall survival analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M. Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols